CLINICAL TRIAL: NCT04366466
Title: Program to Promote Commitment to Care for the Prevention of Suicidal Recurrence (Health Monitoring and Case Management) Versus Usual Treatment (Health Monitoring): Randomized Controlled Interventional Study in Routine Care.
Brief Title: Program to Promote Engagement in Care for the Prevention of Recidivism
Acronym: PEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Januel (Other)
Responsible Party: Sponsor-Investigator, Januel, Head of clinical research unit, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10477M-PEPS
Record Dates: First submitted 2020-04-16; First posted 2020-04-29 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Suicide; Health Care Seeking Behavior; Case Management
MeSH Terms: conditions — Suicide; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Controlled, randomized and prospective study of a cohort of suicide victims comparing an experimental (interventional) group to a control group (usual treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suicide attempt patient who will receive sanitory supervision (Other): The control group will establish the health monitoring
  Interventions: Other: suicide attempt patient using PEPS Program
- Suicide attempt patient who will participate to PEPS Program (Experimental): The intervention group will test the program of Promotion of Commitment to Care for the Prevention of Suicidal Recidivism.
  Interventions: Other: suicide attempt patient using PEPS Program

INTERVENTIONS:
Other: suicide attempt patient using PEPS Program — The research protocol consists of two phases separated by randomization.
  A Hospital Phase common to both groups:
  Day zero is the day of the suicide attempt for which the patient came to the hospital.
  A post-hospital phase including the P.E.P.S. program for the intervention group and telephone reminders for the usual treatment group.
  Other Names: Suicide attempt patient using sanitary supervision

SUMMARY:
In France, the number of emergency visits for suicide attempts is estimated at 220,000 per year. Suicide management aims to reduce suicide risk factors in order to improve the mental health of patients and prevent recurrences.

To day, no study has compared the approaches to health surveillance and case management in a clinical trial, nor established the benefit of each on commitment to care and beyond the prevention of suicidal recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18.
* Male and female.
* Admission to CH St Denis for a suicide attempt.
* Referral for outpatient follow-up.
* Patient with no psychiatric follow-up or who has been out of follow-up for at least three months.
* Patient having given their written informed consent.

Exclusion Criteria:

* Patients not affiliated with social security or state medical aid.
* Patients who do not have the required faculties to be evaluated (cognitive and delusional disorders).
* Patients treated for more than 72 hours after their procedure (maximum length of stay in the UAS and/or in medical intensive care.
* Patient currently under psychiatric care.
* Patients who cannot be called back by telephone (no telephone, homeless, incarceration).
* Patients who do not master the French language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) | Day 0
  rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders.
Suicide Intent Scale | Day 0
  The Suicide Intent Scale (SIS) developed by A.T. BECK in 1974, is the only scale that focuses solely on the assessment of the suicide attempt that has just taken place.
Montgomery-Asberg depression rating scale | Day 0
  This scale is widely used to measure the changes brought about by the treatment of depression. It assesses the severity of symptoms in a wide variety of areas such as mood, sleep and appetite, physical and mental fatigue, and thoughts of suicide.

SECONDARY OUTCOMES:
Evaluating the effectiveness of the P.E.P.S. program in preventing suicidal recidivism | 1 year
  percentage of all suicidants who relapse during the 12-month study period.
Evaluate the level of possible generalization of the program | 1 year
  percentage of all suicides of subjects likely to benefit from the program (subjects fulfilling the inclusion and non-inclusion criteria).
Evaluate the feasibility of the program | 1 year
  percentage of subjects included in the intervention group who received all interventions); weighted by the percentage of acceptance to participate in the study

CONTACTS AND LOCATIONS:
Overall Officials: Fayçal MOUAFFAK, Principal Investigator — Investigateur Principal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617